CLINICAL TRIAL: NCT01441934
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Effect of Sildenafil in the Treatment of Patients With Pulmonary Hypertension Associated to Chronic Obstructive Lung Disease
Brief Title: SPHERIC-1. Sildenafil and Pulmonary HypERtension In COPD
Acronym: SPHERIC-1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Italian Association of Hospital Pneumologists (Other)
Responsible Party: Principal Investigator, Dr. Patrizio Vitulo, Head of Pulmonary Medicine, The Mediterranean Institute for Transplantation and Advanced Specialized Therapies
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARC209
Record Dates: First submitted 2011-07-29; First posted 2011-09-28 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: Pulmonary Hypertension; COPD
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil citrate (Active Comparator): 20 mg t.i.d.
  Interventions: Drug: Sildenafil citrate
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Sugar pills

INTERVENTIONS:
Drug: Sildenafil citrate — sildenafil 20 mg t.i.d. compared to placebo 20 mg t.i.d - 16 weeks treatment
  Other Names: Revatio
  Arms: Sildenafil citrate
Drug: Sugar pills — placebo t.i.d.
  Arms: Sugar pill

SUMMARY:
Although pulmonary hypertension (PH) is a quite frequent complication of advanced pulmonary diseases, and it is an independent prognostic factor, until now no evidence-based treatment approach exists for those patients.

This study will address if the drug sildenafil can lower pulmonary vascular resistance in patients with significant pulmonary hypertension (high blood pressure in the lungs) associated to chronic obstructive pulmonary disease (COPD). It will see if this treatment can improve effort capacity, quality of life without causing a deterioration in pulmonary gas exchange (mainly arterial oxygenation).

Patients 18 years of age and older with moderate COPD and pulmonary hypertension (mean pulmonary arterial pressure >30 mmHg) may be eligible for this study. Participants are randomly assigned to receive sildenafil or placebo (pill with no drug) for 16 weeks.

Before starting treatment (baseline), and a the end of the study, the patients have a comprehensive assessment including:

* a chest x-ray and CT scan (only at baseline);
* pulmonary function tests to measure how much air the patient can breathe in and out, and the capacity of diffusion of gases;
* arterial blood gases analysis (for safety reason this examination is performed at baseline, before the randomization after one hour from the administration of a tablet (20 mg) of sildenafil, and every month)
* an echocardiogram (heart ultrasound) (only at baseline);
* a 6-minute walk test to measure exercise capacity;
* a quality-of-life assessment (SF-36 questionnaire)
* a right heart catheterization to evaluate the severity of hypertension

At the end of the 16-week period, patients may opt to continue to receive sildenafil and monitoring in an open-label phase of the study for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patient affected by stable COPD under optimal treatment, chronic oxygen therapy in patients with hypoxia, with PaO2 at rest ≥ 60 mmHg and PaCO2≤ 55 mmHg, aged between 18 and 80 years old:
* Group 1: BPCO GOLD I-III (post bronchodilator FEV1 ≥ 30%, FEV1/FVC ≤ 0,7 , TLC ≥ 70%) + PAPm ≥ 30 mmHg and PCP <15 mmHg
* Group 2: BPCO GOLD IV (post bronchodilator FEV1 <30%, FEV1/FVC ≤ 0,7 , TLC ≥ 70%) + PAPm ≥ 35 mmHg and PCP <15 mmHg

Exclusion Criteria:

* Different types of pulmonary hypertension (chronic, thromboembolic pulmonary hypertension, pulmonary arterial hypertension etc.)
* Significant left cardiac disease (LVEF <45%, cardiomyopathy, valvulopathy, unstable coronaropathy)
* Treatment with nitrates in the last 10 days, or in need of other nitrate therapy for different diseases
* Treatment with other specific drugs for arterial pulmonary hypertension (less than 4 weeks)
* Significant systemic disease other than COPD
* Recent exacerbations of chronic bronchitis (< 4 weeks)
* Pregnancy or breastfeeding, or women without an adequate contraceptive method for the whole study duration
* History of anaphylaxis or allergic reactions to 5-phosphodiesterase inhibitors
* Cancers within the last 5 years with the exception of localized cancers of the skin or of the cervix
* Hepatic insufficiency or chronic renal failure or hemoglobinemia < 10 g/dL during the screening phase
* Contraindications to subministration as per SPC
* Mental disorder, alcohol abuse, chronic alcoholism, drug abuse
* Subjects unable to sign the informed consent form
* Subjects unable to walk

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Pulmonary vascular resistance (PVR) | 16 weeks
  PVR are measured by right cath study as the following formula:
  PVR= (mean pulmonary arterial pressure-pulmonary arterial wedge pressure)/cardiac output

SECONDARY OUTCOMES:
Arterial blood gas analysis | 16 Weeks
Pulmonary function - Borg scale | 16 Weeks
  The dyspnea is assessed by an analogic scale from 0 (no dyspnea) to 10 (very severe dyspnea)
Pulmonary function - Bode Index | 16 Weeks
  The BODE Index is a composite marker of disease taking into consideration the systemic nature of COPD: FEV1% pred = predicted amount as a percentage of the forced expiratory lung volume in one second; 6MWD = six minute walking distance; MMRC = modified medical research council dyspnea scale; BMI = body mass index.
Functional capacity - Quality of Life | 16 Weeks
  Quality of Life is assessed by a standardized questionnaire (SF-36 questionnaire) at baseline and the end of study
Functional capacity testing - 6 Minutes walking test | 16 Weeks
  The six-minute walk test is performed in a straight corridor (length 25-30 meters) in the same environmental conditions

CONTACTS AND LOCATIONS:
Overall Officials: Patrizio Vitulo, MD, Study Chair — Dept. of Medicine - Pulmonary Medicine - IsMeTT Palermo, Italy; Carmine D. Vizza, MD, Study Chair — Pulmonary Hypertension Center - Dept. of Cardiovascular and Respiratory Sciences - I° School of Medicine - Sapienza University of Rome (Italy)
Locations (10):
- Italy (10):
  - Pulmonary Unit - Azienda Ospedaliera Ospedale Niguarda Ca' Granda, Milan, Milano
  - Pulmonary Diseases Clinic - Azienda Ospedaliera Universitaria - Policlinico di Modena, Modena, Modena
  - Pulmonary Clinic - Federico II University - Azienda Ospedaliera V. Monaldi, Napoli, Napoli
  - Thoracic Surgery Clinic - Azienda Ospedaliera di Padova, Padua, Padova
  - Dept. of Medicine - Pulmonary Medicine - IsMeTT, Palermo, Palermo
  - Pulmonary Diseases Clinic - Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia
  - Pulmonary Hypertension Center - Policlinico Umberto I, Rome, Rome
  - University Pulmonary Unit - Azienda Ospedaliera Universitaria Senese, Siena, Siena
  - Pulmonary Unit - Azienda Ospedaliera Universitaria San Giovanni Battista, Torino, Torino
  - Pulmonary Unit - Azienda Ospedaliera Universitaria Ospedali Riuniti di Trieste, Trieste, Trieste